CLINICAL TRIAL: NCT00577967
Title: Gabapentin - A Solution to Uremic Pruritus? A Prospective, Randomized, Placebo-controlled, Double-blind Study
Brief Title: Gabapentin - A Solution to Uremic Pruritus?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 355/05; HARECCTR0500020
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Pruritus; Uremia
Keywords: Uremic pruritis
MeSH Terms: conditions — Pruritus; Uremia | interventions — Gabapentin

INTERVENTIONS:
Drug: Gabapentin

SUMMARY:
To investigate using the drug gabapentin to relieve the intense pruritic sensation associated with chronic renal failure patients undergoing peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese male and female patients aged > 18 undergoing CAPD for at least 3 months and able to read and understand Chinese
* Patients experiencing moderate to severe pruritis, defined as persistent, treatment-resistant pruritis considerably impairing sleep or daytime activity. Treatment resistance is defined as no or only partial resolvement of pruritis under current anti-pruritis treatment regimens such as anti-pruritis lotions and anti-histamines.
* Patients in stable clinical condition in terms of peritoneal dialysis and general health
* Patients able to understand and answer the SDS questionnaire
* Patients able to express the sensation of itchiness in the terms of the VAS and the SDS score
* Patients who are willing to give written informed consent and to participate in and comply with the study protocol

Exclusion Criteria:

* Patients with a known history of pruritis or dermatologic disease antedating renal failure.
* Patients with skin disease other than the usual cutaneous findings of uraemia such as xerosis or ecchymosis.
* Patients under current treatment with systemic steroids
* Known history of allergy to Gabapentin
* Those patients already put on anti-convulsants
* Unable to give written informed consent for the study
* Pregnancy or female patients of child-bearing age who are unwilling to use contraception
* Poor drug compliance
* Known HIV positivity
* Active neoplastic disease
* Those who do not want to participate the study

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-10; Study Completion 2006-03 (Estimated)

PRIMARY OUTCOMES:
Subjective measurement of reduction in pruritus | 3 months

SECONDARY OUTCOMES:
Tolerability of Gabapentin in CAPD patients | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yui Pong Siu, Dr, Principal Investigator — Medical and Geriatrics / Nephrology, Tuen Mun Hospital
Locations (1):
- Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264